CLINICAL TRIAL: NCT06561503
Title: Evaluation of Health Related Quality of Life in Patients With Intoxication-type Inherited Metabolic Diseases in Sohag University Hospital
Status: Recruiting | Type: Observational
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Alaa Mahmoud Aly, Resident-pediatric department-sohag hospital university, Sohag University
Other Study IDs: Soh-Med-24-07-16MS
Record Dates: First submitted 2024-08-12; First posted 2024-08-20 (Actual); Last update posted 2024-08-20 (Actual); Status verified 2024-08

CONDITIONS: Intoxication-type Inherited Metabolic Diseases

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- cases group: Metabolic Cases

SUMMARY:
Intoxication-type Inherited Metabolic disease (IT-IMD) are a group of rare, chronic diseases. They share the pattern of intoxication by a substance, which accumulates due to a genetically determined enzyme failure. In many IT-IMD, brain toxicity is predominant. Treatment mostly encompasses a lifelong natural protein-restricted diet, supplementation of amino acid solutions and specific medication.(1) The diseases are by definition chronic but according to their characteristics they can be subdivided into having or having not acute, crisis-like episodes. Patients with ITIMD such as urea cycle disorders (UCD) or organic acidurias (OA) may be challenged by life-threatening metabolic crises and acute exacerbations (acute IT-IMD). Many acute IT-IMD patients develop neurocognitive and behavioural problems, often despite sufficient treatment adherence. Furthermore, difficulties to adhere to diet and medication, nausea and vomiting are major every-day complaints.(2) Phenylketonuria (PKU), an inborn error of phenylalanine (Phe) metabolism is a non-acute IT-IMD, patients generally have no metabolic crises or short-term disease exacerbations. Accumulating Phe is toxic to the brain and causes severe, irreversible cognitive impairment. Mainstay of treatment in classical PKU is a lifelong protein-restricted diet complemented with amino acid supplementation.(3)With good metabolic control, classical PKU patients usually achieve normal cognitive functioning, but complaints such as attention problems, anxiety, or depression occur frequently.(2) Acute and non-acute IT-IMD patients face considerable burdens of disease and treatment, which may impair health-related quality of life (HrQoL). HrQoL is 'a patient's perception of the impact of disease and treatment on functioning in a variety of dimensions, including physical, psychological, and social domains.(1,4) Research on the subjective burden of IT-IMD remains sparse. . Previous research suggests that pediatric patients' and their parents' everyday life is significantly affected by the considerable disease and treatment burdens of E-IMD.(5) Studies with appropriate sample sizes are needed to make valid statements about health-related quality of life (HrQoL) in children and adolescents with IT-IMD

DETAILED DESCRIPTION:
Type of the study:

Prospective observational study.

Place of the study:

Metabolic and Genetic Unit, Department of Pediatrics, Faculty of Medicine, Sohag University, Sohag, Egypt.

Inclusion Criteria:

* Confirmed diagnosis of PKU(chronic and acute crisis(, gluatric acidemia, methylmalonic acidemia, Isovaleric academia and Propionic academia.
* Patients and their parents agree to participate in the study. Exclusion Criteria:.
* Patients and their parents refuse to participate in the study.
* Children with incomplete medical records or unavailable clinical data.
* Non diagnosed cases.

Study duration:

One year (starting from obtaining approval from the research ethics committee).

Patients:

Our study will include all children diagnosed with IT-IMD at the Metabolic and Genetic Unit of Sohag University

ELIGIBILITY:
Inclusion Criteria:

* • Confirmed diagnosis of PKU(chronic and acute crisis(, gluatric acidemia, methylmalonic acidemia, Isovaleric academia and Propionic academia.

  * Patients and their parents agree to participate in the study

Exclusion Criteria:

* Patients and their parents refuse to participate in the study.

  * Children with incomplete medical records or unavailable clinical data.
  * Non diagnosed cases.

Ages: 1 Day to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: - • Confirmed diagnosis of PKU(chronic and acute crisis(, gluatric acidemia, methylmalonic acidemia, Isovaleric academia and Propionic academia.
  • Patients and their parents agree to participate in the study
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2024-08-01 (Actual); Primary Completion 2025-08-01 (Estimated); Study Completion 2025-08-01 (Estimated)

PRIMARY OUTCOMES:
Health-related quality of life (HrQoL) questionnaire | 1 year
  quality of life in patients with Intoxication-type Inherited Metabolic Diseases

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag university Hospital, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Zeltner NA, Baumgartner MR, Bondarenko A, Ensenauer R, Karall D, Kolker S, Muhlhausen C, Scholl-Burgi S, Thimm E, Quitmann J, Burgard P, Landolt MA, Huemer M. Development and Psychometric Evaluation of the MetabQoL 1.0: A Quality of Life Questionnaire for Paediatric Patients with Intoxication-Type Inborn Errors of Metabolism. JIMD Rep. 2017;37:27-35. doi: 10.1007/8904_2017_11. Epub 2017 Mar 1. PMID 28247338
- [Background] Villani GR, Gallo G, Scolamiero E, Salvatore F, Ruoppolo M. "Classical organic acidurias": diagnosis and pathogenesis. Clin Exp Med. 2017 Aug;17(3):305-323. doi: 10.1007/s10238-016-0435-0. Epub 2016 Sep 9. PMID 27613073
- [Background] Varni JW, Seid M, Rode CA. The PedsQL: measurement model for the pediatric quality of life inventory. Med Care. 1999 Feb;37(2):126-39. doi: 10.1097/00005650-199902000-00003. PMID 10024117
- [Background] van Spronsen FJ, van Wegberg AM, Ahring K, Belanger-Quintana A, Blau N, Bosch AM, Burlina A, Campistol J, Feillet F, Gizewska M, Huijbregts SC, Kearney S, Leuzzi V, Maillot F, Muntau AC, Trefz FK, van Rijn M, Walter JH, MacDonald A. Key European guidelines for the diagnosis and management of patients with phenylketonuria. Lancet Diabetes Endocrinol. 2017 Sep;5(9):743-756. doi: 10.1016/S2213-8587(16)30320-5. Epub 2017 Jan 10. PMID 28082082